CLINICAL TRIAL: NCT03907488
Title: A Phase III, Randomized Study of Nivolumab (Opdivo) Plus AVD or Brentuximab Vedotin (Adcetris) Plus AVD in Patients (Age >/= 12 Years) With Newly Diagnosed Advanced Stage Classical Hodgkin Lymphoma
Brief Title: Immunotherapy (Nivolumab or Brentuximab Vedotin) Plus Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage III-IV Classic Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01960; NCI-2019-01960 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1826 (Other: SWOG); S1826 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Ann Arbor Stage III Hodgkin Lymphoma; Ann Arbor Stage III Lymphocyte-Depleted Classic Hodgkin Lymphoma; Ann Arbor Stage III Mixed Cellularity Classic Hodgkin Lymphoma; Ann Arbor Stage III Nodular Sclerosis Classic Hodgkin Lymphoma; Ann Arbor Stage IV Hodgkin Lymphoma; Ann Arbor Stage IV Lymphocyte-Depleted Classic Hodgkin Lymphoma; Ann Arbor Stage IV Mixed Cellularity Classic Hodgkin Lymphoma; Ann Arbor Stage IV Nodular Sclerosis Classic Hodgkin Lymphoma; Classic Hodgkin Lymphoma; Lymphocyte-Rich Classic Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Specimen Handling; Brentuximab Vedotin; Dacarbazine; Doxorubicin; Filgrastim; Granulocyte Colony-Stimulating Factor; Magnetic Resonance Spectroscopy; Nivolumab; pegfilgrastim; pegylated granulocyte colony-stimulating factor; Radiotherapy; Radiation; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (chemotherapy, nivolumab, radiation) (Experimental): Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, dacarbazine IV, and nivolumab IV over 30 minutes on days 1 and 15. Patients may receive pegfilgrastim SC on days 2 and 16, or filgrastim SC or IV on days 6-10 and 21-25. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 6, patients may receive radiation therapy 5 days per week for approximately 4 weeks at the discretion of the treating physician. Patients also undergo peripheral blood specimen collection and CT, PET/CT and MRI on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Biological: Filgrastim; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Biological: Pegfilgrastim; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Vinblastine Sulfate
- Arm II (chemotherapy, brentuximab vedotin, radiation) (Experimental): Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, dacarbazine IV, and brentuximab vedotin IV over 30 minutes on days 1 and 15. Patients may receive pegfilgrastim SC on days 2 and 16, or filgrastim SC or IV on days 6-10 and 21-25. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 6, patients may receive radiation therapy 5 days per week for approximately 4 weeks at the discretion of the treating physician. Patients also undergo peripheral blood specimen collection and CT, PET/CT and MRI on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Brentuximab Vedotin; Procedure: Computed Tomography; Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Biological: Filgrastim; Procedure: Magnetic Resonance Imaging; Biological: Pegfilgrastim; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy; Drug: Vinblastine Sulfate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo peripheral blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN 35; SGN-35; SGN35
  Arms: Arm II (chemotherapy, brentuximab vedotin, radiation)
Procedure: Computed Tomography — Undergo PET/CT or CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; FI106; hydroxydaunorubicin; Rubex
Biological: Filgrastim — Given SC or IV
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Filgrastim Biosimilar Tbo-filgrastim; Filgrastim XM02; Filgrastim-aafi; Filgrastim-ayow; Filgrastim-sndz; G-CSF; Granix; Neupogen; Neutroval; Nivestim; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; Releuko; rG-CSF; Tbo-filgrastim; Tevagrastim; XM02; Zarxio
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm I (chemotherapy, nivolumab, radiation)
Biological: Pegfilgrastim — Given SC
  Other Names: Dulastin; Filgrastim SD-01; filgrastim-SD/01; Fulphila; Fylnetra; G-Lasta; HSP-130; Jinyouli; Neulasta; Neulastim; Neupopeg; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; Pegfilgrastim-apgf; Pegfilgrastim-bmez; Pegfilgrastim-cbqv; Pegfilgrastim-fpgk; Pegfilgrastim-jmdb; Pegfilgrastim-pbbk; Pegylated G-CSF; Pegylated GCSF; Pegylated Granulocyte Colony Stimulating Factor; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Stimufend; Tripegfilgrastim; Udenyca; Ziextenzo
Procedure: Positron Emission Tomography — Undergo PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Receive radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Vinblastine Sulfate — Given IV
  Other Names: 29060 LE; 29060-LE; Exal; Velban; Velbe; Velsar; VINCALEUKOBLASTINE

SUMMARY:
This phase III trial compares immunotherapy drugs (nivolumab or brentuximab vedotin) when given with combination chemotherapy in treating patients with newly diagnosed stage III or IV classic Hodgkin lymphoma. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Brentuximab vedotin is a monoclonal antibody, brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to cancer cells in a targeted way and delivers vedotin to kill them. Chemotherapy drugs, such as doxorubicin, vinblastine, and dacarbazine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. The addition of nivolumab or brentuximab vedotin to combination chemotherapy may shrink the cancer or extend the time without disease symptoms coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the progression-free survival (PFS) in patients with newly diagnosed advanced stage classical Hodgkin lymphoma randomized to N-AVD (nivolumab, doxorubicin hydrochloride [doxorubicin], vinblastine sulfate [vinblastine], dacarbazine) versus that obtained with BV-AVD (brentuximab vedotin, doxorubicin, vinblastine, dacarbazine).

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) in patients randomized to N-AVD versus BV-AVD.

II. To compare event-free survival (EFS) in patients randomized to N-AVD versus BV-AVD.

III. To compare the metabolic complete response (CR) rate at the end of treatment in patients randomized to N-AVD versus BV-AVD.

IV. To compare the physician-reported treatment-related adverse event rates between arms stratified by age groups.

V. To compare patient-reported symptoms using selected Patient Reported Outcome Common Toxicity Criteria for Adverse Events (PRO-CTCAE) items between arms stratified by age groups.

VI. To compare the safety and tolerability of N-AVD versus that of BV-AVD.

QUALITY OF LIFE OBJECTIVE:

I. To compare between arms patient-reported fatigue, neuropathy and health-related quality of life over time (baseline, beginning of cycle 3, 4-8 weeks after the last dose of protocol therapy [following last dose of study drug or radiation therapy, whichever is later], and 1 and 3 years after randomization) using the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue, the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx), and the PROMIS Global, respectively.

BANKING OBJECTIVES:

I. To bank specimens for future correlative studies. II. To bank positron emission tomography (PET)-computed tomography (CT) images for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive doxorubicin hydrochloride intravenously (IV), vinblastine sulfate IV, dacarbazine IV, and nivolumab IV over 30 minutes on days 1 and 15. Patients may receive pegfilgrastim subcutaneously (SC) on days 2 and 16, or filgrastim SC or IV on days 6-10 and 21-25. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 6, patients may receive radiation therapy 5 days per week for approximately 4 weeks at the discretion of the treating physician. Patients also undergo peripheral blood specimen collection and CT, PET/CT and/or magnetic resonance imaging (MRI) on study.

ARM II: Patients receive doxorubicin hydrochloride IV, vinblastine sulfate IV, dacarbazine IV, and brentuximab vedotin IV over 30 minutes on days 1 and 15. Patients may receive pegfilgrastim SC on days 2 and 16, or filgrastim SC or IV on days 6-10 and 21-25. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 6, patients may receive radiation therapy 5 days per week for approximately 4 weeks at the discretion of the treating physician. Patients also undergo peripheral blood specimen collection and CT, PET/CT and MRI on study.

After completion of study treatment and prior to disease progression, patients are followed up every 3 months for the first year, every 6 months for years 2 and 3, then annually until 10 years after registration. Patients are followed up at the time of progression and then annually until 10 years after registration. Patients who receive radiation therapy are followed up at 8-12 weeks after completion of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically confirmed newly diagnosed, previously untreated stage III or IV classical Hodgkin lymphoma (nodular sclerosing, mixed cellularity, lymphocyte-rich, or lymphocyte-depleted, or not otherwise specified [NOS]). Nodular lymphocyte predominant Hodgkin lymphoma is not eligible.
* Patients must have bidimensionally measurable disease (at least one lesion with longest diameter >= 1.5 cm) documented on the Lymphoma Baseline Tumor Assessment Form in Rave.
* Patients must have a whole body or limited whole body PET-CT scan performed within 42 days prior to registration. (A contrast-enhanced [diagnostic] CT, MRI or MR-PET is acceptable in event that PET-CT is contra-indicated, however if it is later possible to administer a PET-CT, then PET-CT is strongly preferred for the interim scan (after cycle 2) (if performed) and the EOT assessment. Otherwise, if PET-CT is not subsequently possible, then the same modality as baseline must be used throughout the trial.) NOTE: All images from PET-CT, CT, MRI or MR-PET scans performed as standard of care to assess disease (within 42 days prior to registration) must be submitted and associated radiology reports must be submitted.
* Patients must be >= 12 years of age.
* Patients must not have received any prior chemotherapy, radiation, or antibody-based treatment for classical Hodgkin lymphoma. Steroid pre-treatment is permitted.
* Patients must not have had prior solid organ transplant.
* Patients must not have had prior allogeneic stem cell transplantation.
* Patients must not have received a live vaccine within 30 days prior to planned day 1 of protocol therapy (e.g. measles, mumps, rubella, varicella, yellow fever, rabies, Bacillus Calmette-Guerin [BCG], oral polio vaccine, and oral typhoid).
* At registration, investigator must declare intent-to-treat with residual PET radiation therapy (residual PET RT- RPRT) to be administered after patient completes 6 cycles of therapy if, after end of treatment, the patient meets criteria specified for receiving RT). Patients will be stratified by investigator's intent-to-treat with residual PET RT.

  * All pediatric patients (< 18 years of age) will be considered intent-to-treat with Residual PET RT at time of registration.
* Patients must have a performance status corresponding to Zubrod scores of 0, 1 or 2. Use Lansky for patients =< 17 years of age. *The conversion of the Lansky to Eastern Cooperative Oncology Group (ECOG) scales is intended for National Cancer Institute (NCI) reporting purposes only.
* Adults (age 18 or older): Creatinine clearance >= 30 mL/min, as estimated by the Cockcroft and Gault formula. The creatinine value used in the calculation must have been obtained within 28 days prior to registration. Estimated creatinine clearance is based on actual body weight.

Pediatric Patients (age 12-17), the following must have been obtained within 14 days prior to registration:

* Measured or calculated creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2, or
* Serum creatinine =< 1.5 x institutional upper limit of normal (IULN), or a serum creatinine (SCr) based on age/gender as follows:

  * Age < 13 maximum serum creatinine: Male 1.2 mg/dL; Female 1.2 mg/dL
  * Age 13 to < 16 maximum serum creatinine: Male 1.5 mg/dL; Female 1.4 mg/dL
  * Age 16-17 maximum serum creatinine: Male 1.7 mg/dL; Female 1.4 mg/dL

    * Total bilirubin =< 2 x IULN (must be documented within 28 days prior to registration for adults [age 18 or older]; must be documented within 14 days prior to registration for pediatric patients [age 12-17]).
* Unless due to Gilbert's disease, lymphomatous involvement of liver or vanishing bile duct syndrome

  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x IULN (must be documented within 28 days prior to registration for adults [age 18 or older]; must be documented within 14 days prior to registration for pediatric patients [age 12-17]).
* Unless due to Gilbert's disease, lymphomatous involvement of liver or vanishing bile duct syndrome

  * Patients must have an echocardiogram (ECHO), multigated acquisition (MUGA), or functional cardiac imaging scan with a left ventricular ejection (LVEF) fraction >= 50% or a shortening fraction of >= 27%. For all patients, the ECHO, MUGA, or functional cardiac imaging scan must be performed within 42 days prior to registration.
  * Patients with known human immunodeficiency virus (HIV) infection must be receiving anti-retroviral therapy and have an undetectable or unquantifiable viral load at their most recent viral load test within 6 months prior to registration.
  * Patients must not have known active hepatitis B (HBV) or hepatitis C virus (HCV) at date of registration. Patients with previously treated HBV or HCV that have an undetectable viral load within 6 months prior to registration and no residual hepatic impairment are eligible.
  * Patients must not have any known central nervous system lymphoma.
  * Patients must not have a history of or active interstitial pneumonitis or interstitial lung disease.
  * Patients must not have had a diagnosis of inherited or acquired immunodeficiency.
  * Patients must not have any known uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, hemodynamically unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
  * Patients must not have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to registration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Steroid use for the control of Hodgkin lymphoma symptoms is allowable, but must be discontinued prior to cycle 1, day 1.
  * Patients with peripheral neuropathy must have < grade 2 at date of registration.
  * Patients must not have active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, immunosuppressive drugs, or corticosteroids with doses higher than prednisone 10 mg or equivalent). Autoimmune diseases include but are not limited to autoimmune hepatitis, inflammatory bowel disease (including ulcerative colitis and Crohn's disease), as well as symptomatic disease (e.g.: rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); central nervous system (CNS) or motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis, multiple sclerosis or glomerulonephritis). Vitiligo, alopecia, hypothyroidism on stable doses of thyroid replacement therapy, psoriasis not requiring systemic therapy within the past 2 years are permitted.
  * No second prior malignancy is allowed except for adequately treated basal (or squamous cell) skin cancer, any in situ cancer or other cancer for which the patient has been disease free for two years.
  * Females of childbearing potential must not be pregnant or nursing, and have a negative pregnancy test within 28 days prior to registration. Women/men of reproductive potential must have agreed to use an effective contraceptive method while receiving study drug and for women until 6 months after receiving the last dose of study drug or, for men, until 7 months after receiving the last dose of study drug. A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures.
  * Patients must have one formalin-fixed paraffin embedded (FFPE) diagnostic tumor block or at least 1 diagnostic, 4-5 micron, hematoxylin and eosin (H&E) slide collected prior to registration and available for submission.
  * Patients must be offered participation in banking for planned translational medicine and future research. With patient consent, any residuals from the mandatory tissue submission will also be banked for future research.
  * Patients who can complete Patient-Reported Outcome instruments in English, Spanish, or French must complete the PROMIS Fatigue, the FACT/GOG-Ntx, and the PROMIS Global prior to registration. Patients who do not complete PRO instruments prior to registration but are otherwise eligible will remain eligible for the primary analysis and other secondary analyses.
  * Patients who can complete Patient-Reported Outcome instruments in English, Spanish, or French must also agree to complete the PROMIS Fatigue, the FACT/GOG-Ntx, the PROMIS Global, and the PRO-CTCAE (or Pediatric [Ped] PRO-CTCAE) at the scheduled on-study assessment timepoints.
  * Patients must be informed of the investigational nature of this study and all patients and/or their parents or legal guardians (for patients < 18 years of age) must sign and give informed consent and assent (where appropriate) in accordance with institutional and federal guidelines. For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board Initiative (CIRB) regulations.
* Note: As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 994 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2026-03-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — SWOG Cancer Research Network
Locations (731):
- United States (714):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Children's Hospital of Orange County, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Palms West Radiation Therapy, Loxahatchee Groves, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - UChicago Medicine AdventHealth Cancer Institute Hinsdale, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Children's Hospital-Park Ridge, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - STCC at DHR Health Institute for Research and Development, Edinburg, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Valley Medical Center, Renton, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (15):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - William Osler Health System-Brampton Civic Hospital, Brampton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CHA Hopital L'Enfant-Jesus, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec
- Puerto Rico (2):
  - HIMA San Pablo Oncologic Hospital, Caguas
  - University Pediatric Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Herrera AF, LeBlanc M, Castellino SM, Li H, Rutherford SC, Evens AM, Davison K, Punnett A, Parsons SK, Ahmed S, Casulo C, Bartlett NL, Tuscano JM, Mei MG, Hess BT, Jacobs R, Saeed H, Torka P, Hu B, Moskowitz C, Kaur S, Goyal G, Forlenza C, Doan A, Lamble A, Kumar P, Chowdhury S, Brinker B, Sharma N, Singh A, Blum KA, Perry AM, Kovach AE, Hodgson D, Constine LS, Shields LK, Prica A, Dillon H, Little RF, Shipp MA, Crump M, Kahl B, Leonard JP, Smith SM, Song JY, Kelly KM, Friedberg JW. Nivolumab+AVD in Advanced-Stage Classic Hodgkin's Lymphoma. N Engl J Med. 2024 Oct 17;391(15):1379-1389. doi: 10.1056/NEJMoa2405888. PMID 39413375
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Chemotherapy, Nivolumab, Radiation) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation)
Started | 496 | 498
Completed | 450 | 425
Not Completed | 46 | 73
Not completed — Adverse Event | 20 | 20
Not completed — Withdrawal by Subject | 9 | 13
Not completed — Lack of Efficacy | 0 | 9
Not completed — Death | 3 | 8
Not completed — not protocol specified | 5 | 8
Not completed — Ineligible | 9 | 15

BASELINE CHARACTERISTICS:
Population: Modified intent to treat group, in participants deemed ineligible are excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Chemotherapy, Nivolumab, Radiation) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation) | Total
Number analyzed (Participants) | 487 | 483 | 970
Age, Continuous [Median (Full Range); unit: years] | 27.6 [12.0 to 83.7] | 26.8 [12.0 to 81.7] | 27 [12.0 to 83.7]
Age, Customized [Count of Participants; unit: Participants]
  Age, Stratified: 12-17 | 118 | 118 | 236
  Age, Stratified: 18-60 | 321 | 318 | 639
  Age, Stratified: >60 | 48 | 47 | 95
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 210 | 426
  Male | 271 | 273 | 544
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 372 | 361 | 733
  Black | 58 | 56 | 114
  Asian | 11 | 17 | 28
  Other or unknown | 46 | 49 | 95
  Hispanic | 66 | 58 | 124

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Will be reported as the number of participants who have experienced death or progression, measured at two years. Progression will be measured according to the 2014 Lugano classification. Will test the null hypothesis (HR=1) for PFS using stratified log-rank test with a one-sided alpha of 0.021. The analysis will be based on modified intent-to-treat and will include all eligible patients as randomized regardless of treatment received. The one-sided alpha of .021 will control of the overall type-one error of the study (including the 2 interim superiority analyses) to be less than .025.
Time Frame: From date of registration to date of first observation of progressive disease, or death due to any cause, assessed at 2 years
Population: All the patients who underwent randomization except for those who were deemed to be ineligible by pathology review or owing to violation of the eligibility criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chemotherapy, Nivolumab, Radiation) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation)
Number analyzed (Participants) | 487 | 483
Participants | 41 | 81
Statistical Analysis 1: Comparison: Arm I (Chemotherapy, Nivolumab, Radiation) vs Arm II (Chemotherapy, Brentuximab Vedotin, Radiation); The primary analysis of PFS used a stratified log rank test statistic and is reported as two-sided test. Stratified Cox regression was used to estimate treatment hazard ratios for treatment effect. 95% two-sided intervals are reported. The Kaplan-Meier method was used to estimate PFS curves; Test type: Superiority; p < 0.005, Log Rank — One sided P-value

2. Secondary Outcome: Overall Survival
Description: Will be reported as the count of participants who have died, measured at two years. Stratified log-rank test at two-sided alpha level of .05.
Time Frame: From date of registration to two years or death.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chemotherapy, Nivolumab, Radiation) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation)
Number analyzed (Participants) | 487 | 483
Participants | 7 | 14

3. Secondary Outcome: Event-free Survival (EFS)
Description: Will be reported as count of participants who have experienced an EFS event or death at two years.
  EFS Events are defined as:
  * Disease progression/relapse
  * Administration of non-protocol specified systemic anti-lymphoma therapy (i.e. salvage therapy) at any time after initiation of protocol therapy.
  * Administration of any non-protocol specified radiation therapy at any time afterinitiation of protocol therapy Will be estimated using Kaplan-Meier method and compared between treatment arms using cox regression model.
Time Frame: From date of registration to date of first occurrence of EFS event, assessed at 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chemotherapy, Nivolumab, Radiation) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation)
Number analyzed (Participants) | 487 | 483
Participants | 52 | 91

4. Secondary Outcome: Number of Participants With of Adverse Events
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Chemotherapy, Nivolumab, Radiation) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation)
Number analyzed (Participants) | 481 | 476
Participants
  Abdominal distension | 1 | 3
  Abdominal pain | 61 | 110
  Activated partial thromboplastin time prolonged | 2 | 3
  Acute kidney injury | 3 | 3
  Adrenal insufficiency | 2 | 0
  Agitation | 4 | 0
  Akathisia | 1 | 0
  Alanine aminotransferase increased | 163 | 209
  Alkaline phosphatase increased | 58 | 84
  Allergic reaction | 4 | 6
  Allergic rhinitis | 0 | 3
  Alopecia | 103 | 127
  Amenorrhea | 1 | 5
  Amnesia | 1 | 0
  Anal fissure | 0 | 1
  Anal fistula | 0 | 1
  Anal hemorrhage | 1 | 1
  Anemia | 198 | 222
  Anorectal infection | 1 | 0
  Anorexia | 61 | 107
  Anosmia | 3 | 1
  Anxiety | 20 | 30
  Appendicitis | 1 | 0
  Arthralgia | 65 | 60
  Arthritis | 3 | 0
  Ascites | 1 | 0
  Aspartate aminotransferase increased | 129 | 168
  Ataxia | 0 | 3
  Atelectasis | 1 | 1
  Atrial fibrillation | 1 | 1
  Autoimmune disorder | 1 | 0
  Back pain | 27 | 35
  Bacteremia | 0 | 2
  Belching | 3 | 1
  Bladder infection | 1 | 1
  Bloating | 7 | 18
  Blood and lymphatic system disorders - Other, spec | 3 | 5
  Blood bicarbonate decreased | 3 | 5
  Blood bilirubin increased | 14 | 14
  Blood lactate dehydrogenase increased | 18 | 25
  Blurred vision | 11 | 15
  Bone pain | 41 | 99
  Brachial plexopathy | 0 | 1
  Breast pain | 0 | 1
  Bronchial infection | 2 | 0
  Bronchospasm | 1 | 0
  Bruising | 2 | 8
  Bullous dermatitis | 0 | 1
  Burn | 0 | 1
  Buttock pain | 1 | 0
  CD4 lymphocytes decreased | 0 | 1
  CPK increased | 1 | 1
  Cardiac arrest | 0 | 2
  Cardiac disorders - Other, specify | 6 | 0
  Cardiac troponin I increased | 1 | 0
  Cardiac troponin T increased | 1 | 0
  Catheter related infection | 1 | 3
  Cheilitis | 1 | 0
  Chest pain - cardiac | 4 | 0
  Chest wall pain | 2 | 1
  Chills | 22 | 20
  Cholesterol high | 0 | 1
  Chronic kidney disease | 1 | 0
  Cognitive disturbance | 3 | 0
  Colitis | 6 | 6
  Colonic obstruction | 0 | 1
  Concentration impairment | 4 | 7
  Confusion | 3 | 2
  Conjunctivitis | 1 | 4
  Conjunctivitis infective | 0 | 2
  Constipation | 196 | 209
  Cough | 33 | 32
  Creatinine increased | 27 | 13
  Cyanosis | 1 | 0
  Dehydration | 14 | 32
  Delirium | 0 | 1
  Depressed level of consciousness | 1 | 2
  Depression | 10 | 10
  Dermatitis radiation | 0 | 2
  Diarrhea | 101 | 130
  Disseminated intravascular coagulation | 1 | 0
  Dizziness | 29 | 40
  Dry eye | 2 | 3
  Dry mouth | 19 | 32
  Dry skin | 15 | 17
  Dysarthria | 1 | 0
  Dysesthesia | 0 | 3
  Dysgeusia | 37 | 60
  Dysmenorrhea | 1 | 0
  Dyspepsia | 34 | 21
  Dysphagia | 8 | 7
  Dysphasia | 0 | 1
  Dyspnea | 43 | 58
  Dysuria | 3 | 1
  Ear and labyrinth disorders - Other, specify | 1 | 0
  Ear pain | 0 | 1
  Eczema | 3 | 7
  Edema face | 1 | 5
  Edema limbs | 17 | 17
  Ejection fraction decreased | 3 | 3
  Electrocardiogram QT corrected interval prolonged | 1 | 0
  Electrocardiogram T wave abnormal | 1 | 0
  Endocrine disorders - Other, specify | 9 | 0
  Enterocolitis | 2 | 1
  Enterocolitis infectious | 1 | 4
  Eosinophilia | 12 | 16
  Epistaxis | 10 | 16
  Erectile dysfunction | 2 | 0
  Erythema multiforme | 1 | 1
  Erythroderma | 1 | 0
  Esophageal pain | 1 | 0
  Esophagitis | 2 | 3
  Extrapyramidal disorder | 1 | 2
  Eye disorders - Other, specify | 3 | 3
  Facial muscle weakness | 1 | 0
  Facial pain | 1 | 4
  Fall | 5 | 9
  Fatigue | 232 | 246
  Febrile neutropenia | 28 | 33
  Fecal incontinence | 0 | 1
  Fever | 64 | 63
  Fibrinogen decreased | 2 | 0
  Flank pain | 1 | 3
  Flashing lights | 1 | 1
  Flatulence | 4 | 6
  Floaters | 0 | 1
  Flu like symptoms | 4 | 3
  Flushing | 10 | 3
  Folliculitis | 2 | 2
  Fracture | 0 | 1
  GGT increased | 4 | 4
  Gait disturbance | 0 | 2
  Gastric hemorrhage | 0 | 1
  Gastritis | 9 | 8
  Gastroesophageal reflux disease | 27 | 40
  Gastrointestinal disorders - Other, specify | 10 | 14
  Gastrointestinal pain | 1 | 0
  Gastroparesis | 0 | 1
  General disorders and administration site conditio | 7 | 6
  Generalized edema | 1 | 0
  Generalized muscle weakness | 16 | 25
  Glucose intolerance | 1 | 0
  Glucosuria | 2 | 2
  Guillain-Barre syndrome | 0 | 1
  Gynecomastia | 0 | 1
  Headache | 71 | 77
  Heart failure | 2 | 1
  Hematuria | 4 | 0
  Hemolysis | 1 | 0
  Hemorrhoidal hemorrhage | 1 | 0
  Hemorrhoids | 4 | 1
  Hepatic failure | 2 | 0
  Hepatobiliary disorders - Other, specify | 2 | 1
  Herpes simplex reactivation | 1 | 3
  Hiccups | 6 | 11
  Hoarseness | 0 | 4
  Hot flashes | 9 | 20
  Hypercalcemia | 6 | 10
  Hyperglycemia | 57 | 67
  Hyperhidrosis | 14 | 16
  Hyperkalemia | 5 | 4
  Hyperlipidemia | 0 | 1
  Hypermagnesemia | 4 | 3
  Hypernatremia | 1 | 5
  Hyperphosphatemia | 17 | 16
  Hypertension | 41 | 43
  Hyperthyroidism | 13 | 0
  Hypertriglyceridemia | 2 | 2
  Hyperuricemia | 6 | 9
  Hypoalbuminemia | 43 | 41
  Hypocalcemia | 34 | 35
  Hypoglycemia | 7 | 6
  Hypokalemia | 31 | 64
  Hypomagnesemia | 5 | 22
  Hyponatremia | 30 | 57
  Hypoparathyroidism | 1 | 0
  Hypophosphatemia | 11 | 19
  Hypotension | 18 | 18
  Hypothyroidism | 36 | 3
  Hypoxia | 3 | 3
  INR increased | 3 | 1
  Ileus | 0 | 4
  Immune system disorders - Other, specify | 1 | 1
  Infections and infestations - Other, specify | 18 | 12
  Infusion related reaction | 36 | 10
  Infusion site extravasation | 2 | 2
  Injection site reaction | 1 | 2
  Injury, poisoning and procedural complications - O | 1 | 0
  Insomnia | 30 | 54
  Investigations - Other, specify | 13 | 10
  Irregular menstruation | 4 | 5
  Irritability | 1 | 1
  Joint range of motion decreased | 0 | 2
  Laryngopharyngeal dysesthesia | 1 | 0
  Lethargy | 3 | 2
  Leukocytosis | 2 | 6
  Libido decreased | 6 | 3
  Lip infection | 3 | 0
  Lipase increased | 2 | 1
  Localized edema | 3 | 3
  Lung infection | 10 | 14
  Lymph gland infection | 1 | 0
  Lymph node pain | 1 | 3
  Lymphocyte count decreased | 109 | 114
  Lymphocyte count increased | 4 | 10
  Malaise | 8 | 3
  Memory impairment | 8 | 4
  Menorrhagia | 1 | 1
  Metabolism and nutrition disorders - Other, specif | 5 | 2
  Mitral valve disease | 1 | 0
  Movements involuntary | 1 | 2
  Mucosal infection | 1 | 1
  Mucositis oral | 109 | 100
  Muscle cramp | 14 | 19
  Muscle weakness lower limb | 5 | 7
  Muscle weakness trunk | 1 | 0
  Muscle weakness upper limb | 1 | 2
  Musculoskeletal and connective tissue disorder - | 5 | 6
  Myalgia | 54 | 58
  Myositis | 2 | 0
  Nail changes | 2 | 9
  Nail discoloration | 7 | 16
  Nail infection | 3 | 2
  Nail ridging | 1 | 1
  Nasal congestion | 6 | 12
  Nausea | 317 | 331
  Neck edema | 3 | 2
  Neck pain | 4 | 3
  Neoplasms benign, malignant and unspecified (incl | 2 | 0
  Nervous system disorders - Other, specify | 5 | 8
  Neuralgia | 2 | 3
  Neutrophil count decreased | 275 | 166
  Non-cardiac chest pain | 16 | 16
  Oral dysesthesia | 6 | 6
  Oral hemorrhage | 0 | 1
  Oral pain | 30 | 24
  Pain | 43 | 31
  Pain in extremity | 22 | 36
  Palmar-plantar erythrodysesthesia syndrome | 1 | 2
  Palpitations | 7 | 2
  Pancreatic enzymes decreased | 0 | 1
  Pancreatitis | 4 | 1
  Papulopustular rash | 4 | 3
  Paresthesia | 36 | 43
  Paronychia | 1 | 2
  Paroxysmal atrial tachycardia | 2 | 0
  Pelvic pain | 1 | 2
  Penile infection | 0 | 1
  Pericardial effusion | 1 | 0
  Pericarditis | 3 | 0
  Peripheral motor neuropathy | 21 | 36
  Peripheral sensory neuropathy | 141 | 268
  Pharyngeal mucositis | 1 | 0
  Pharyngitis | 0 | 1
  Phlebitis | 3 | 4
  Photophobia | 1 | 2
  Photosensitivity | 1 | 2
  Platelet count decreased | 53 | 89
  Pleural effusion | 2 | 1
  Pleuritic pain | 1 | 0
  Pneumonitis | 11 | 15
  Postnasal drip | 2 | 1
  Presyncope | 2 | 3
  Productive cough | 2 | 2
  Proteinuria | 2 | 2
  Pruritus | 48 | 25
  Psychiatric disorders - Other, specify | 1 | 3
  Psychosis | 0 | 1
  Pulmonary edema | 1 | 1
  Rash acneiform | 16 | 12
  Rash maculo-papular | 55 | 59
  Rash pustular | 0 | 1
  Rectal fissure | 0 | 1
  Rectal hemorrhage | 1 | 2
  Rectal pain | 1 | 4
  Renal and urinary disorders - Other, specify | 1 | 1
  Respiratory failure | 0 | 3
  Respiratory, thoracic and mediastinal disorders - | 3 | 6
  Restrictive cardiomyopathy | 1 | 0
  Rhabdomyolysis | 1 | 0
  Rhinorrhea | 6 | 8
  Salivary duct inflammation | 1 | 2
  Scalp pain | 1 | 0
  Scrotal pain | 0 | 1
  Seizure | 2 | 1
  Sepsis | 8 | 15
  Serum amylase increased | 1 | 0
  Sinus bradycardia | 1 | 3
  Sinus disorder | 0 | 1
  Sinus tachycardia | 17 | 25
  Skin and subcutaneous tissue disorders - Other, sp | 16 | 18
  Skin hyperpigmentation | 8 | 8
  Skin hypopigmentation | 3 | 0
  Skin infection | 6 | 10
  Skin ulceration | 0 | 1
  Small intestinal obstruction | 0 | 1
  Sneezing | 0 | 1
  Somnolence | 0 | 1
  Sore throat | 16 | 27
  Spasticity | 1 | 1
  Stomach pain | 10 | 10
  Stroke | 1 | 0
  Superficial thrombophlebitis | 3 | 3
  Supraventricular tachycardia | 0 | 1
  Syncope | 1 | 2
  Tendon reflex decreased | 1 | 1
  Testicular pain | 0 | 2
  Thromboembolic event | 12 | 10
  Thrush | 7 | 14
  Thyroid stimulating hormone increased | 28 | 1
  Tinnitus | 8 | 6
  Tooth discoloration | 0 | 1
  Tooth infection | 1 | 0
  Toothache | 3 | 2
  Tracheal mucositis | 0 | 1
  Tracheitis | 1 | 0
  Tremor | 4 | 3
  Tumor lysis syndrome | 1 | 1
  Tumor pain | 0 | 1
  Typhlitis | 0 | 3
  Upper gastrointestinal hemorrhage | 1 | 0
  Upper respiratory infection | 7 | 8
  Urinary frequency | 2 | 2
  Urinary incontinence | 1 | 1
  Urinary retention | 0 | 1
  Urinary tract infection | 7 | 12
  Urinary tract pain | 2 | 0
  Urinary urgency | 0 | 1
  Urticaria | 1 | 2
  Vaginal discharge | 2 | 0
  Vaginal infection | 2 | 4
  Vascular access complication | 1 | 2
  Vascular disorders - Other, specify | 3 | 1
  Vasovagal reaction | 0 | 1
  Ventricular arrhythmia | 1 | 1
  Ventricular tachycardia | 1 | 1
  Vertigo | 2 | 1
  Vision decreased | 3 | 0
  Voice alteration | 1 | 2
  Vomiting | 138 | 160
  Watering eyes | 1 | 5
  Weight gain | 13 | 8
  Weight loss | 25 | 71
  Wheezing | 2 | 1
  White blood cell decreased | 202 | 136
  Wound infection | 0 | 1

5. Secondary Outcome: Metabolic Complete Response Rate
Description: This outcome measure will be reported by 11/5/2025.
Time Frame: 4-8 weeks after last dose of study drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Adverse events will be assessed using CTCAE version 5.0. All cause mortality will be reported as all cause mortality within the two year time frame that was analyzed for the primary endpoint.
  Please note that the number of participants at risk for all-cause mortality is greater than the number of participants at risk for adverse events. Only participants who received intervention are eligible for adverse events reporting.
Arm/Group | Arm I (Chemotherapy, Nivolumab, Radiation) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation)
All-Cause Mortality (participants affected / at risk) | 7/487 | 14/483
Serious Adverse Events (participants affected / at risk) | 140/481 | 18/476
Other Adverse Events (participants affected / at risk) | 468/481 | 465/476
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy, Nivolumab, Radiation) (N=481) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation) (N=476)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Blood and lymphatic system disorders-Other (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 4
Hemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac disorders-Other (Cardiac disorders) | 2 | 0
Chest pain - cardiac (Cardiac disorders) | 4 | 0
Heart failure (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0
Pericarditis (Cardiac disorders) | 3 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 6 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 2
Chills (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Edema limbs (General disorders) | 1 | 0
Fever (General disorders) | 10 | 0
Generalized edema (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Allergic reaction (Immune system disorders) | 3 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 18 | 0
Lung infection (Infections and infestations) | 5 | 1
Sepsis (Infections and infestations) | 11 | 6
Skin infection (Infections and infestations) | 2 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Cardiac troponin T increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
GGT increased (Investigations) | 1 | 0
INR increased (Investigations) | 3 | 0
Investigations-Other (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 30 | 3
Platelet count decreased (Investigations) | 7 | 1
White blood cell decreased (Investigations) | 11 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Lethargy (Nervous system disorders) | 1 | 0
Nervous system disorders-Other (Nervous system disorders) | 4 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pregnancy, puerperium and perinatal conditions-Oth (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Confusion (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Hematuria (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory, thoracic and mediastinal disorders-Ot (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 1
Thromboembolic event (Vascular disorders) | 10 | 0
Vascular disorders-Other (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Chemotherapy, Nivolumab, Radiation) (N=481) | Arm II (Chemotherapy, Brentuximab Vedotin, Radiation) (N=476)
Anemia (Blood and lymphatic system disorders) | 251 | 252
Eosinophilia (Blood and lymphatic system disorders) | 23 | 28
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 30
Sinus tachycardia (Cardiac disorders) | 46 | 71
Hypothyroidism (Endocrine disorders) | 38 | 3
Blurred vision (Eye disorders) | 28 | 24
Abdominal pain (Gastrointestinal disorders) | 93 | 164
Bloating (Gastrointestinal disorders) | 13 | 27
Constipation (Gastrointestinal disorders) | 238 | 240
Diarrhea (Gastrointestinal disorders) | 130 | 173
Dry mouth (Gastrointestinal disorders) | 26 | 38
Dyspepsia (Gastrointestinal disorders) | 49 | 33
Gastroesophageal reflux disease (Gastrointestinal disorders) | 47 | 54
Mucositis oral (Gastrointestinal disorders) | 120 | 108
Nausea (Gastrointestinal disorders) | 338 | 354
Oral pain (Gastrointestinal disorders) | 37 | 27
Vomiting (Gastrointestinal disorders) | 156 | 182
Chills (General disorders) | 32 | 29
Edema limbs (General disorders) | 33 | 33
Fatigue (General disorders) | 283 | 277
Fever (General disorders) | 96 | 99
Non-cardiac chest pain (General disorders) | 47 | 42
Pain (General disorders) | 72 | 70
Infections and infestations-Other (Infections and infestations) | 62 | 71
Upper respiratory infection (Infections and infestations) | 21 | 25
Infusion related reaction (Injury, poisoning and procedural complications) | 39 | 16
Alanine aminotransferase increased (Investigations) | 180 | 232
Alkaline phosphatase increased (Investigations) | 85 | 109
Aspartate aminotransferase increased (Investigations) | 148 | 187
Blood lactate dehydrogenase increased (Investigations) | 29 | 39
Creatinine increased (Investigations) | 42 | 23
Lymphocyte count decreased (Investigations) | 123 | 126
Neutrophil count decreased (Investigations) | 277 | 171
Platelet count decreased (Investigations) | 55 | 92
Thyroid stimulating hormone increased (Investigations) | 30 | 6
Weight gain (Investigations) | 52 | 33
Weight loss (Investigations) | 45 | 88
White blood cell decreased (Investigations) | 206 | 141
Anorexia (Metabolism and nutrition disorders) | 78 | 122
Dehydration (Metabolism and nutrition disorders) | 16 | 45
Hyperglycemia (Metabolism and nutrition disorders) | 141 | 148
Hyperphosphatemia (Metabolism and nutrition disorders) | 33 | 30
Hypoalbuminemia (Metabolism and nutrition disorders) | 85 | 77
Hypocalcemia (Metabolism and nutrition disorders) | 63 | 59
Hypokalemia (Metabolism and nutrition disorders) | 50 | 96
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 40
Hyponatremia (Metabolism and nutrition disorders) | 58 | 98
Hypophosphatemia (Metabolism and nutrition disorders) | 17 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 89 | 79
Back pain (Musculoskeletal and connective tissue disorders) | 65 | 78
Bone pain (Musculoskeletal and connective tissue disorders) | 71 | 138
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 18 | 34
Muscle cramp (Musculoskeletal and connective tissue disorders) | 28 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 76 | 79
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 | 71
Dizziness (Nervous system disorders) | 55 | 64
Dysgeusia (Nervous system disorders) | 48 | 65
Headache (Nervous system disorders) | 110 | 123
Paresthesia (Nervous system disorders) | 43 | 46
Peripheral motor neuropathy (Nervous system disorders) | 25 | 38
Peripheral sensory neuropathy (Nervous system disorders) | 158 | 280
Anxiety (Psychiatric disorders) | 95 | 101
Depression (Psychiatric disorders) | 35 | 35
Insomnia (Psychiatric disorders) | 82 | 108
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 21 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 118 | 108
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 96 | 109
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23 | 28
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 34 | 42
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 27 | 44
Sore throat (Respiratory, thoracic and mediastinal disorders) | 40 | 56
Alopecia (Skin and subcutaneous tissue disorders) | 108 | 136
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 34
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 37 | 55
Pruritus (Skin and subcutaneous tissue disorders) | 84 | 67
Rash acneiform (Skin and subcutaneous tissue disorders) | 26 | 34
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 84 | 94
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 42 | 39
Hot flashes (Vascular disorders) | 27 | 32
Hypertension (Vascular disorders) | 79 | 83
Hypotension (Vascular disorders) | 18 | 33

LIMITATIONS AND CAVEATS:
Our trial has several limitations, including the short follow-up time. Secondary analyses and subgroup analyses that involved specified stratification factors were preplanned, but these analyses did not have adequate statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03907488/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03907488/ICF_002.pdf